CLINICAL TRIAL: NCT01555294
Title: Evaluation of Non-invasive Measurements of Atherosclerosis in Cardiovascular Risk Stratification: a Study in a Population-based Cohort and Familial Combined Hyperlipidemia
Brief Title: Evaluation of Non-invasive Measurements of Atherosclerosis in Cardiovascular Risk Stratification
Acronym: NIMA
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Jacqueline de Graaf, Prof. Dr. J. de Graaf, Radboud University Medical Center
Other Study IDs: CMO 2003/174
Record Dates: First submitted 2011-09-06; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Cardiovascular Disease
Keywords: (subclinical)atherosclerosis; non-invasive measurements; intima-media thickness; flow-mediated dilation; pulse wave velocity and analysis; fatal and non-fatal cardiovascular events; ankle-brachial index (at rest and after exercise); general population; Familial Combined Hyperlipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Hyperlipidemia, Familial Combined

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- community-based cohort: The present study is a substudy in the Nijmegen Biomedical Study (NBS). The NBS is a prospective population survey aimed at investigating the frequency of genetic variations in the general population. The study population is recruited as a sex- and age-stratified random sample of all inhabitants of Nijmegen 20 to 90 years old (n=10.000). Recruitment has started in october 2001.
  In the current study 1517 participants aged 50-70 years were included from 2005 to 2008, from whom baseline characteristics were obtained. All visited our hospital and during the visit venous blood was drawn, height and weight were measured, a questionnaire about medical history, life style habits, and family history was completed and non-invasive measurements of atherosclerosis were performed.
- Familial Combined Hyperlipidemia: FCH is the most common inherited dyslipidemia in man. Affected individuals are characterized by elevated cholesterol and/or triglyceride levels and an increased risk of CVD. Our data base contains a unique population of 40 well-characterized FCH families, including 687 patients, relatives and spouses. These families were recruited in 1994 and extensively studied, including information on an extensive panel of biochemical and genetic parameters. In total 343 participants were included in the NIMA study; 103 FCH patients and 240 unaffected relatives from whom baseline characteristics were obtained.

SUMMARY:
Multiple risk factors contribute to atherosclerosis, which ultimately results in clinical manifestation of cardiovascular disease. Atherosclerosis results in both functional and morphological changes in the vessel wall, which can be measured by ultrasonography. The current study has been designed to

1. To evaluate whether non-invasive measurements of atherosclerosis are independent predictors of cardiovascular disease and
2. to delineate new biochemical parameters and genetic variations, allowing earlier and more effective preventive therapy
3. The investigators intend to set guidelines for use of NIMA in an outpatient setting to facilitate early detection of increased cardiovascular risk and monitor life-style and pharmaceutical interventions.

In both the general population and in Familial Combined Hyperlipidemia.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the major cause of death in all developed countries. Atherosclerosis is the main cause of CVD. Abundant evidence indicates the 4 major independent risk factors for atherosclerosis and CVD include cigarette smoking, elevated blood pressure, elevated total cholesterol and diabetes mellitus. However, a major problem in clinical medicine is that at every level of risk factor exposure, there is a large inter-individual variation in the amount of atherosclerosis and the development of CVD. Therefore, it is difficult to predict the CVD risk in an individual patient based on risk factor screening alone.

Non-invasive measurements of atherosclerosis (NIMA): An indicator of the overall effect of all known and unknown potential risk factors for atherosclerosis in vivo can be assessed by measuring atherosclerosis directly in the vessel wall. This also provides the opportunity to measure atherosclerosis before developing symptoms of CVD, as changes in the arterial wall precede clinical symptoms of CVD.

Objectives: (1)The main objective is to evaluate whether NIMA are independent predictors of CVD and thus add information to traditional risk factor stratification. (2) Furthermore, we will delineate new biochemical and genetic risk factors, allowing earlier and more effective preventive therapy. (3) We intend to set guidelines for use of NIMA in an outpatient setting to facilitate early detection of increased cardiovascular risk and monitor life-style and pharmaceutical interventions.

We will evaluate 4 different NIMA, based on ultrasound and tonometry techniques, including intima media thickness (IMT), endothelial function by flow mediated dilation (FMD), ankle-brachial index (ABI), Pulse Wave Analyses(PWA) and pulse wave velocity (PWV). The power of NIMA, to predict cardiovascular events will be studied in two available populations, a low risk population cohort, the Nijmegen Biomedical Study (NBS) and a high risk population, families with Familial Combined Hyperlipidemia.

The NBS is a prospective population survey aimed at investigating the frequency of genetic variations in the general population. The study population is recruited as a sex- and age-stratified random sample of all inhabitants of Nijmegen 20 to 90 years old (n=10.000). Recruitment has started in October 2001. The present study is a substudy in the NBS. A follow-up approach will be used to evaluate whether NIMA are related to future cardiovascular events. In total 1517 participants aged 50-70 years were included.

FCH is the most common inherited hyperlipidemia in man. Affected individuals are characterized by elevated cholesterol and/or triglyceride levels and other associated traits including small-dense LDL, insulin resistance, oxidative stress and increased apoB levels, which have been proposed to contribute to the increased risk of CVD. So, this population will be most informative to evaluate the relevance of NIMA in CVD risk assessment as patients exhibit numerous, additive risk factors, which are missed in traditional cardiovascular risk assessment. Our data base contains a unique population of 40 well-characterized FCH families, including 687 patients, relatives and spouses with 5 years follow-up data. These families participate in an ongoing long-term follow-up program with registration of CVD.

All four NIMA's, including IMT, ABI, PWV/PWA, FMD, and both traditional and new biochemical and genetic parameters will be measured in both populations. The relevance of NIMA in identifying subjects at increased risk of CVD will be determined. Furthermore, the effect of risk factors on IMT, ABI, PWV and FMD will be studied, including clinical and traditional risk factors and new biochemical parameters and genetic variations.

Innovative aspects: We will develop an evidence based protocol for NIMA to show the presence of atherosclerosis before clinical manifestation of CVD and to improve cardiovascular risk stratification beyond traditional risk factor screening. Furthermore, we will delineate new risk factors, including both biochemical parameters and genetic variations, contributing to design optimal (new) treatment and to develop new strategies for prevention of CVD in the general population and in a high risk population, FCH.

Clinical relevance: If NIMA turns out to provide powerful information in identifying subjects at increased risk of CVD we will incorporate NIMA into clinical practice guidelines for the purpose of cardiovascular risk stratification and evaluation of risk management strategies. The identification of potential new biochemical and/or genetic risk factors will be very helpful to design optimal treatment and to develop new strategies for identification and prevention of CVD in both the general population and families with FCH.

ELIGIBILITY:
Population-based cohort:

Inclusion Criteria:

* aged 50-70 years at inclusion

Exclusion Criteria:

* recent symptomatic CV disease (<6 months)

Familial Combined Hyperlipidemia:

Inclusion Criteria:

* age >18 years

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants recruited from a population-based survey aged 50-70 years. Participants from families with Familial Combined Hyperlipidemia.
Sampling Method: Non-Probability Sample
Enrollment: 1960 (Actual)
Dates: Start 2005-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Cardiovascular events | 3-7 years
  Fatal and non-fatal cardiovascular events will be evaluated by questionnaire and validated using hospital records and records from general practitioners.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline de Graaf, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, Dept. of General Internal Medicine, Division of Vascular Medicine; Anton FH Stalenhoef, MD, PhD, Study Chair — Radboud University Nijmegen Medical Centre, Dept. of General Internal Medicine, Division of Vascular Medicine; Martin den Heijer, MD, PhD, Study Chair — Radboud University Nijmegen Medical Centre, Dept. of Epidemiology and Biostatistics; Suzanne Holewijn, PhD, Study Chair — Radboud University Nijmegen Medical Centre, Dept. of General Internal Medicine, Division of Vascular Medicine
Locations (1):
- Radboud University Nijmegen Medical Centre, Department of General Internal Medicine, Division of Vascular Medicine, Nijmegen, Netherlands

REFERENCES:
- [Background] Gretarsdottir S, Baas AF, Thorleifsson G, Holm H, den Heijer M, de Vries JP, Kranendonk SE, Zeebregts CJ, van Sterkenburg SM, Geelkerken RH, van Rij AM, Williams MJ, Boll AP, Kostic JP, Jonasdottir A, Jonasdottir A, Walters GB, Masson G, Sulem P, Saemundsdottir J, Mouy M, Magnusson KP, Tromp G, Elmore JR, Sakalihasan N, Limet R, Defraigne JO, Ferrell RE, Ronkainen A, Ruigrok YM, Wijmenga C, Grobbee DE, Shah SH, Granger CB, Quyyumi AA, Vaccarino V, Patel RS, Zafari AM, Levey AI, Austin H, Girelli D, Pignatti PF, Olivieri O, Martinelli N, Malerba G, Trabetti E, Becker LC, Becker DM, Reilly MP, Rader DJ, Mueller T, Dieplinger B, Haltmayer M, Urbonavicius S, Lindblad B, Gottsater A, Gaetani E, Pola R, Wells P, Rodger M, Forgie M, Langlois N, Corral J, Vicente V, Fontcuberta J, Espana F, Grarup N, Jorgensen T, Witte DR, Hansen T, Pedersen O, Aben KK, de Graaf J, Holewijn S, Folkersen L, Franco-Cereceda A, Eriksson P, Collier DA, Stefansson H, Steinthorsdottir V, Rafnar T, Valdimarsson EM, Magnadottir HB, Sveinbjornsdottir S, Olafsson I, Magnusson MK, Palmason R, Haraldsdottir V, Andersen K, Onundarson PT, Thorgeirsson G, Kiemeney LA, Powell JT, Carey DJ, Kuivaniemi H, Lindholt JS, Jones GT, Kong A, Blankensteijn JD, Matthiasson SE, Thorsteinsdottir U, Stefansson K. Genome-wide association study identifies a sequence variant within the DAB2IP gene conferring susceptibility to abdominal aortic aneurysm. Nat Genet. 2010 Aug;42(8):692-7. doi: 10.1038/ng.622. Epub 2010 Jul 11. PMID 20622881
- [Result] ter Avest E, Holewijn S, Stalenhoef AF, de Graaf J. Variation in non-invasive measurements of vascular function in healthy volunteers during daytime. Clin Sci (Lond). 2005 May;108(5):425-31. doi: 10.1042/CS20040300. PMID 15636580
- [Result] ter Avest E, Abbink EJ, Holewijn S, de Graaf J, Tack CJ, Stalenhoef AF. Effects of rosuvastatin on endothelial function in patients with familial combined hyperlipidaemia (FCH). Curr Med Res Opin. 2005 Sep;21(9):1469-76. doi: 10.1185/030079905X61910. PMID 16197666
- [Result] ter Avest E, Holewijn S, Bredie SJ, Stalenhoef AF, de Graaf J. Remnant particles are the major determinant of an increased intima media thickness in patients with familial combined hyperlipidemia (FCH). Atherosclerosis. 2007 Mar;191(1):220-6. doi: 10.1016/j.atherosclerosis.2006.03.025. Epub 2006 May 4. PMID 16677651
- [Result] ter Avest E, Holewijn S, Bredie SJ, van Tits LJ, Stalenhoef AF, de Graaf J. Pulse wave velocity in familial combined hyperlipidemia. Am J Hypertens. 2007 Mar;20(3):263-9. doi: 10.1016/j.amjhyper.2006.09.015. PMID 17324737
- [Result] Ter Avest E, Holewijn S, van Tits LJ, de Wit HM, Stalenhoef AF, de Graaf J. Endothelial function in familial combined hyperlipidaemia. Eur J Clin Invest. 2007 May;37(5):381-9. doi: 10.1111/j.1365-2362.2007.01804.x. PMID 17461984
- [Result] Koenen TB, van Tits LJ, Holewijn S, Lemmers HL, den Heijer M, Stalenhoef AF, de Graaf J. Adiponectin multimer distribution in patients with familial combined hyperlipidemia. Biochem Biophys Res Commun. 2008 Nov 7;376(1):164-8. doi: 10.1016/j.bbrc.2008.08.111. Epub 2008 Aug 30. PMID 18762168
- [Result] Holewijn S, den Heijer M, Swinkels DW, Stalenhoef AF, de Graaf J. The metabolic syndrome and its traits as risk factors for subclinical atherosclerosis. J Clin Endocrinol Metab. 2009 Aug;94(8):2893-9. doi: 10.1210/jc.2009-0084. Epub 2009 May 5. PMID 19417041
- [Result] Holewijn S, den Heijer M, Swinkels DW, Stalenhoef AF, de Graaf J. Brachial artery diameter is related to cardiovascular risk factors and intima-media thickness. Eur J Clin Invest. 2009 Jul;39(7):554-60. doi: 10.1111/j.1365-2362.2009.02152.x. Epub 2009 May 8. PMID 19453648
- [Result] Holewijn S, den Heijer M, van Tits LJ, Swinkels DW, Stalenhoef AF, de Graaf J. Impact of waist circumference versus adiponectin level on subclinical atherosclerosis: a cross-sectional analysis in a sample from the general population. J Intern Med. 2010 Jun;267(6):588-98. doi: 10.1111/j.1365-2796.2009.02192.x. Epub 2009 Nov 4. PMID 20210840
- [Result] Holewijn S, den Heijer M, Swinkels DW, Stalenhoef AF, de Graaf J. Apolipoprotein B, non-HDL cholesterol and LDL cholesterol for identifying individuals at increased cardiovascular risk. J Intern Med. 2010 Dec;268(6):567-77. doi: 10.1111/j.1365-2796.2010.02277.x. PMID 21091808
- [Result] Holewijn S, Sniderman AD, den Heijer M, Swinkels DW, Stalenhoef AF, de Graaf J. Application and validation of a diagnostic algorithm for the atherogenic apoB dyslipoproteinemias: ApoB dyslipoproteinemias in a Dutch population-based study. Eur J Clin Invest. 2011 Apr;41(4):423-33. doi: 10.1111/j.1365-2362.2010.02426.x. Epub 2010 Dec 3. PMID 21128932
- [Result] Bus BA, Marijnissen RM, Holewijn S, Franke B, Purandare N, de Graaf J, den Heijer M, Buitelaar JK, Voshaar RC. Depressive symptom clusters are differentially associated with atherosclerotic disease. Psychol Med. 2011 Jul;41(7):1419-28. doi: 10.1017/S0033291710002151. Epub 2010 Dec 10. PMID 21144110
- [Result] Holewijn S, den Heijer M, Stalenhoef AF, de Graaf J. Non-invasive measurements of atherosclerosis (NIMA): current evidence and future perspectives. Neth J Med. 2010 Dec;68(12):388-99. PMID 21209464
- [Result] Marijnissen RM, Bus BA, Holewijn S, Franke B, Purandare N, de Graaf J, den Heijer M, Buitelaar JK, Oude Voshaar RC. Depressive symptom clusters are differentially associated with general and visceral obesity. J Am Geriatr Soc. 2011 Jan;59(1):67-72. doi: 10.1111/j.1532-5415.2010.03228.x. PMID 21226677
- [Result] Ter Avest E, Stalenhoef AF, de Graaf J. What is the role of non-invasive measurements of atherosclerosis in individual cardiovascular risk prediction? Clin Sci (Lond). 2007 May;112(10):507-16. PMID 17419684
- [Result] de Graaf J, van der Vleuten GM, ter Avest E, Dallinga-Thie GM, Stalenhoef AF. High plasma level of remnant-like particles cholesterol in familial combined hyperlipidemia. J Clin Endocrinol Metab. 2007 Apr;92(4):1269-75. doi: 10.1210/jc.2006-1973. Epub 2007 Jan 16. PMID 17227806
- [Result] van der Vleuten GM, Isaacs A, Zeng WW, ter Avest E, Talmud PJ, Dallinga-Thie GM, van Duijn CM, Stalenhoef AF, de Graaf J. Haplotype analyses of the APOA5 gene in patients with familial combined hyperlipidemia. Biochim Biophys Acta. 2007 Jan;1772(1):81-8. doi: 10.1016/j.bbadis.2006.10.012. Epub 2006 Oct 26. PMID 17157483
- [Result] ter Avest E, Abbink EJ, de Graaf J, Tack CJ, Stalenhoef AF. Effect of rosuvastatin on insulin sensitivity in patients with familial combined hyperlipidaemia. Eur J Clin Invest. 2005 Sep;35(9):558-64. doi: 10.1111/j.1365-2362.2005.01549.x. PMID 16128862
- [Result] Brouwers MC, de Graaf J, van Greevenbroek MM, Georgieva AM, van der Kallen CJ, Ter Avest E, Stehouwer CD, Stalenhoef AF, de Bruin TW. Parabolic relationship between plasma triacylglycerols and LDL-cholesterol in familial combined hyperlipidaemia: the multiple-type hyperlipidaemia explained? Clin Sci (Lond). 2008 Mar;114(5):393-401. doi: 10.1042/CS20070314. PMID 17953518
- [Result] van Himbergen TM, van Tits LJ, Ter Avest E, Roest M, Voorbij HA, de Graaf J, Stalenhoef AF. Paraoxonase (PON1) is associated with familial combined hyperlipidemia. Atherosclerosis. 2008 Jul;199(1):87-94. doi: 10.1016/j.atherosclerosis.2007.10.017. Epub 2007 Dec 21. PMID 18096166
- [Result] Murabito JM, White CC, Kavousi M, Sun YV, Feitosa MF, Nambi V, Lamina C, Schillert A, Coassin S, Bis JC, Broer L, Crawford DC, Franceschini N, Frikke-Schmidt R, Haun M, Holewijn S, Huffman JE, Hwang SJ, Kiechl S, Kollerits B, Montasser ME, Nolte IM, Rudock ME, Senft A, Teumer A, van der Harst P, Vitart V, Waite LL, Wood AR, Wassel CL, Absher DM, Allison MA, Amin N, Arnold A, Asselbergs FW, Aulchenko Y, Bandinelli S, Barbalic M, Boban M, Brown-Gentry K, Couper DJ, Criqui MH, Dehghan A, den Heijer M, Dieplinger B, Ding J, Dorr M, Espinola-Klein C, Felix SB, Ferrucci L, Folsom AR, Fraedrich G, Gibson Q, Goodloe R, Gunjaca G, Haltmayer M, Heiss G, Hofman A, Kieback A, Kiemeney LA, Kolcic I, Kullo IJ, Kritchevsky SB, Lackner KJ, Li X, Lieb W, Lohman K, Meisinger C, Melzer D, Mohler ER 3rd, Mudnic I, Mueller T, Navis G, Oberhollenzer F, Olin JW, O'Connell J, O'Donnell CJ, Palmas W, Penninx BW, Petersmann A, Polasek O, Psaty BM, Rantner B, Rice K, Rivadeneira F, Rotter JI, Seldenrijk A, Stadler M, Summerer M, Tanaka T, Tybjaerg-Hansen A, Uitterlinden AG, van Gilst WH, Vermeulen SH, Wild SH, Wild PS, Willeit J, Zeller T, Zemunik T, Zgaga L, Assimes TL, Blankenberg S, Boerwinkle E, Campbell H, Cooke JP, de Graaf J, Herrington D, Kardia SL, Mitchell BD, Murray A, Munzel T, Newman AB, Oostra BA, Rudan I, Shuldiner AR, Snieder H, van Duijn CM, Volker U, Wright AF, Wichmann HE, Wilson JF, Witteman JC, Liu Y, Hayward C, Borecki IB, Ziegler A, North KE, Cupples LA, Kronenberg F. Association between chromosome 9p21 variants and the ankle-brachial index identified by a meta-analysis of 21 genome-wide association studies. Circ Cardiovasc Genet. 2012 Feb 1;5(1):100-12. doi: 10.1161/CIRCGENETICS.111.961292. Epub 2011 Dec 23. PMID 22199011